CLINICAL TRIAL: NCT01210664
Title: A Phase I Safety Trial of CD4+CD127lo/-CD25+ Polyclonal Treg Adoptive Immunotherapy for the Treatment of Type 1 Diabetes
Brief Title: T1DM Immunotherapy Using CD4+CD127lo/-CD25+ Polyclonal Tregs
Acronym: Treg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSFDC411AI; JDRF4-2005-1168 (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Treg
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyclonal Regulatory T Cells (Experimental): Patients with Type 1 Diabetes Mellitus will have their regulatory T cells (Tregs) isolated by researchers and receive Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells by infusion
  Interventions: Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells

INTERVENTIONS:
Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells — The researchers will multiply/expand the Tregs in the laboratory using anti-CD3/anti-CD28 coated beads plus IL-2. Then, the Tregs will be infused back into the patient in a single infusion. The first cohort will receive 0.05 x10^8 cells. The second cohort will receive 0.4 x10^8 cells. The third cohort will receive 3.2 x10^8 cells. The fourth cohort will receive 26 x10^8 cells.
  Other Names: Tregs

SUMMARY:
The investigational therapy under study in this trial, regulatory T cells (Tregs), offers the hope of stabilizing further destruction of insulin producing beta cells in type 1 diabetes. Tregs are a specialized subset of T cells that function to control the immune response. Pre-clinical studies in non-obese diabetic mice have demonstrated that adoptive transfer of Tregs can slow diabetes progression and, in some cases, reverse new onset diabetes. The primary purpose of this Phase 1 study is to assess the safety and feasibility of intravenous infusion of ex vivo selected and expanded autologous polyclonal Tregs in patients with type 1 diabetes (T1DM) to support dose selection for a future efficacy trial. The study also aims to assess the effect of Tregs on beta cell function as well as on other measures of diabetes severity and the autoimmune response underlying T1DM.

DETAILED DESCRIPTION:
Currently, there is no approved medical treatment for preservation of the body's ability to produce insulin in patients with Type 1 Diabetes Mellitus (T1DM), and the progression of the disease can have devastating consequences. Inadequate blood glucose control results in many long term complications including kidney disease, blindness, amputation and nerve damage. In spite of the advances in insulin therapy and subsequent glucose control, patients are required to infuse insulin subcutaneously daily throughout their lives, monitor their diet and blood sugar levels, and deal with life-long uncertainties. The investigational therapy under study in this trial, regulatory T cells (Tregs), offers the hope of stabilizing diabetes. Tregs are a specialized subset of T cells that function to control the immune response. Pre-clinical studies in non-obese diabetic mice have demonstrated that adoptive transfer of Tregs can slow diabetes progression and, in some cases, reverse new onset diabetes. The primary objective of this study is to assess the safety of a single intravenous infusion of Tregs in patients with T1DM. The study will also assess the effect of Tregs on insulin-producing beta cell function as well as other outcomes related to diabetes management. Researchers will isolate Tregs from the patient's own blood using specific T cell surface markers (CD4, CD25, and CD127). This subset of cells is then expanded in the laboratory by co-stimulating with anti-CD3 and anti-CD28 immobilized on magnetic beads, and with the use of growth medium containing human serum and IL-2. Following the 14-day expansion, anti-CD3/anti-CD28 beads will be removed and the Tregs will be concentrated and consolidated. The cells will then be resuspended in sterile infusion solution at the required concentration and infused back into the patient through a standard peripheral intravenous line. Subjects will be observed overnight in the clinical research center for any possible side effects following the infusion. A total of 14 subjects will be enrolled. The study will involve 4 dosing cohorts with 3 or 4 adults in each cohort. Each cohort will receive increasing amounts of Tregs. Subjects will be followed over five years to assess safety of the Treg therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1DM within >3 and <24 months of screening according to the American Diabetes Association criteria
* Between 18 and 45 years of age
* Positive test for Epstein-Barr antibody
* Positive test for at least one of the following antibodies:

  * ICA512-antibody
  * ICA
  * GAD65-antibody
  * Insulin (if assessed within 10 days of the onset of insulin therapy)
  * ZnT8
* Peak C-peptide >0.1 pmol/ml (>0.3 ng/ml) during MMTT challenge
* Adequate venous access to support draw of 400 ml whole blood and infusion of investigational therapy

Exclusion Criteria:

* Hemoglobin <10.0 g/dL; leukocytes <3,000/µL; neutrophils <1,500/µL; lymphocytes <800/µL; platelets <100,000/µL
* Regulatory T cells present in peripheral blood at <10 per µl as determined by flow cytometry
* Serologic evidence of HIV-1 or HIV-2 infection
* Evidence of current hepatitis B as demonstrated by HBsAg or circulating hepatitis B genomes
* Serologic evidence of hepatitis C infection
* Detectable circulating EBV or CMV genomes or active infection
* Positive PPD skin test defined as greater than or equal to 10 mm induration
* Chronic use of systemic glucocorticoids or other immunosuppressive agents, or biologic immunomodulators within 6 months prior to study entry. Specifically, subjects who have received over 7 days of treatment with 7.5mg of prednisone (or the equivalent) within 6 months prior to study entry will be excluded.
* History of malignancy ( including squamous cell carcinoma of the skin or cervix) except adequately treated basal cell carcinoma
* Any chronic illness or prior treatment which in the opinion of the investigator should preclude participation in the trial
* Pregnant or breastfeeding women, any female who is unwilling to use a reliable and effective form of contraception for 2 years afer Treg dosing and any male who is unwilling to use a reliable and effective form of contraception for 3 months after Treg dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Gitelman, MD, Study Chair — University of California, San Francisco; Jeffrey Bluestone, PhD, Study Director — University of California, San Francisco; Kevan Herold, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Yale University, New Haven, Connecticut

REFERENCES:
- [Background] Chatenoud L, Bluestone JA. CD3-specific antibodies: a portal to the treatment of autoimmunity. Nat Rev Immunol. 2007 Aug;7(8):622-32. doi: 10.1038/nri2134. Epub 2007 Jul 20. PMID 17641665
- [Background] Saudek F, Havrdova T, Boucek P, Karasova L, Novota P, Skibova J. Polyclonal anti-T-cell therapy for type 1 diabetes mellitus of recent onset. Rev Diabet Stud. 2004 Summer;1(2):80-8. doi: 10.1900/RDS.2004.1.80. Epub 2004 Aug 10. PMID 17491669
- [Background] Couri CE, Oliveira MC, Stracieri AB, Moraes DA, Pieroni F, Barros GM, Madeira MI, Malmegrim KC, Foss-Freitas MC, Simoes BP, Martinez EZ, Foss MC, Burt RK, Voltarelli JC. C-peptide levels and insulin independence following autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2009 Apr 15;301(15):1573-9. doi: 10.1001/jama.2009.470. PMID 19366777
- [Background] Tang Q, Bluestone JA. Regulatory T-cell physiology and application to treat autoimmunity. Immunol Rev. 2006 Aug;212:217-37. doi: 10.1111/j.0105-2896.2006.00421.x. PMID 16903917
- [Background] Tang Q, Henriksen KJ, Bi M, Finger EB, Szot G, Ye J, Masteller EL, McDevitt H, Bonyhadi M, Bluestone JA. In vitro-expanded antigen-specific regulatory T cells suppress autoimmune diabetes. J Exp Med. 2004 Jun 7;199(11):1455-65. doi: 10.1084/jem.20040139. PMID 15184499
- [Background] Liu W, Putnam AL, Xu-Yu Z, Szot GL, Lee MR, Zhu S, Gottlieb PA, Kapranov P, Gingeras TR, Fazekas de St Groth B, Clayberger C, Soper DM, Ziegler SF, Bluestone JA. CD127 expression inversely correlates with FoxP3 and suppressive function of human CD4+ T reg cells. J Exp Med. 2006 Jul 10;203(7):1701-11. doi: 10.1084/jem.20060772. Epub 2006 Jul 3. PMID 16818678
- [Background] Putnam AL, Brusko TM, Lee MR, Liu W, Szot GL, Ghosh T, Atkinson MA, Bluestone JA. Expansion of human regulatory T-cells from patients with type 1 diabetes. Diabetes. 2009 Mar;58(3):652-62. doi: 10.2337/db08-1168. Epub 2008 Dec 15. PMID 19074986
- [Background] Levine BL. T lymphocyte engineering ex vivo for cancer and infectious disease. Expert Opin Biol Ther. 2008 Apr;8(4):475-89. doi: 10.1517/14712598.8.4.475. PMID 18352851
- [Background] Rapoport AP, Stadtmauer EA, Aqui N, Vogl D, Chew A, Fang HB, Janofsky S, Yager K, Veloso E, Zheng Z, Milliron T, Westphal S, Cotte J, Huynh H, Cannon A, Yanovich S, Akpek G, Tan M, Virts K, Ruehle K, Harris C, Philip S, Vonderheide RH, Levine BL, June CH. Rapid immune recovery and graft-versus-host disease-like engraftment syndrome following adoptive transfer of Costimulated autologous T cells. Clin Cancer Res. 2009 Jul 1;15(13):4499-507. doi: 10.1158/1078-0432.CCR-09-0418. Epub 2009 Jun 9. PMID 19509133
- [Background] Levine BL, Bernstein WB, Aronson NE, Schlienger K, Cotte J, Perfetto S, Humphries MJ, Ratto-Kim S, Birx DL, Steffens C, Landay A, Carroll RG, June CH. Adoptive transfer of costimulated CD4+ T cells induces expansion of peripheral T cells and decreased CCR5 expression in HIV infection. Nat Med. 2002 Jan;8(1):47-53. doi: 10.1038/nm0102-47. PMID 11786906
- [Background] Miao D, Yu L, Eisenbarth GS. Role of autoantibodies in type 1 diabetes. Front Biosci. 2007 Jan 1;12:1889-98. doi: 10.2741/2195. PMID 17127428
- [Background] Wenzlau JM, Juhl K, Yu L, Moua O, Sarkar SA, Gottlieb P, Rewers M, Eisenbarth GS, Jensen J, Davidson HW, Hutton JC. The cation efflux transporter ZnT8 (Slc30A8) is a major autoantigen in human type 1 diabetes. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17040-5. doi: 10.1073/pnas.0705894104. Epub 2007 Oct 17. PMID 17942684
- [Result] Bluestone JA, Buckner JH, Fitch M, Gitelman SE, Gupta S, Hellerstein MK, Herold KC, Lares A, Lee MR, Li K, Liu W, Long SA, Masiello LM, Nguyen V, Putnam AL, Rieck M, Sayre PH, Tang Q. Type 1 diabetes immunotherapy using polyclonal regulatory T cells. Sci Transl Med. 2015 Nov 25;7(315):315ra189. doi: 10.1126/scitranslmed.aad4134. PMID 26606968
- [Derived] Dong S, Hiam-Galvez KJ, Mowery CT, Herold KC, Gitelman SE, Esensten JH, Liu W, Lares AP, Leinbach AS, Lee M, Nguyen V, Tamaki SJ, Tamaki W, Tamaki CM, Mehdizadeh M, Putnam AL, Spitzer MH, Ye CJ, Tang Q, Bluestone JA. The effect of low-dose IL-2 and Treg adoptive cell therapy in patients with type 1 diabetes. JCI Insight. 2021 Sep 22;6(18):e147474. doi: 10.1172/jci.insight.147474. PMID 34324441
- [Derived] Gitelman SE, Bluestone JA. Regulatory T cell therapy for type 1 diabetes: May the force be with you. J Autoimmun. 2016 Jul;71:78-87. doi: 10.1016/j.jaut.2016.03.011. Epub 2016 Apr 28. PMID 27133597

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyclonal Regulatory T Cells, 0.05 x10^8 Cells: Cohort 1: Patients with Type 1 Diabetes Mellitus will have their regulatory T cells (Tregs) isolated by researchers and receive 0.05 x10^8 cells of Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells by infusion
- Polyclonal Regulatory T Cells, 0.4 x10^8 Cells: Cohort 2: Patients with Type 1 Diabetes Mellitus will have their regulatory T cells (Tregs) isolated by researchers and receive 0.4 x10^8 cells of Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells by infusion
- Polyclonal Regulatory T Cells, 3.2 x10^8 Cells: Cohort 3: Patients with Type 1 Diabetes Mellitus will have their regulatory T cells (Tregs) isolated by researchers and receive 3.2 x10^8 cells of Ex vivo expanded Human Autologous Polyclonal Regulatory T Cells by infusion
- Polyclonal Regulatory T Cells, 26 x10^8 Cells: Cohort 4: Patients with Type 1 Diabetes Mellitus will have their regulatory T cells (Tregs) isolated by researchers and receive 26 x10^8 cells of Ex vivo expanded Human Autologous Polyclonal Regulatory T Cells by infusion
Period: Cohort 1: PolyTregs 0.05 x 10^8 Cells
Arm/Group | Polyclonal Regulatory T Cells, 0.05 x10^8 Cells | Polyclonal Regulatory T Cells, 0.4 x10^8 Cells | Polyclonal Regulatory T Cells, 3.2 x10^8 Cells | Polyclonal Regulatory T Cells, 26 x10^8 Cells
Started | 3 | 0 | 0 | 0
Received Study Treatment | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2: PolyTregs 0.4 x 10^8 Cells
Arm/Group | Polyclonal Regulatory T Cells, 0.05 x10^8 Cells | Polyclonal Regulatory T Cells, 0.4 x10^8 Cells | Polyclonal Regulatory T Cells, 3.2 x10^8 Cells | Polyclonal Regulatory T Cells, 26 x10^8 Cells
Started | 0 | 3 | 0 | 0
Received Study Treatment | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3: PolyTregs 3.2 x 10^8 Cells
Arm/Group | Polyclonal Regulatory T Cells, 0.05 x10^8 Cells | Polyclonal Regulatory T Cells, 0.4 x10^8 Cells | Polyclonal Regulatory T Cells, 3.2 x10^8 Cells | Polyclonal Regulatory T Cells, 26 x10^8 Cells
Started | 0 | 0 | 5 | 0
Received Study Treatment | 0 | 0 | 4 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Treg Manufacturing Failure | 0 | 0 | 1 | 0
Period: Cohort 4: PolyTregs 26 x 10^8 Cells
Arm/Group | Polyclonal Regulatory T Cells, 0.05 x10^8 Cells | Polyclonal Regulatory T Cells, 0.4 x10^8 Cells | Polyclonal Regulatory T Cells, 3.2 x10^8 Cells | Polyclonal Regulatory T Cells, 26 x10^8 Cells
Started | 0 | 0 | 0 | 5
Received Study Treatment | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Treg Manufacturing Failure | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants treated with single infusion of PolyTregs
Arm/Group | Polyclonal Regulatory T Cells
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: The number of AEs are reported by cohort and severity.
Time Frame: Mean follow-up of 31 months
Population: Safety analysis includes 14 treated participants who received one dose of PolyTregs at Day 0, two participants who underwent blood draw but did not receive PolyTregs were also included in the safety analysis.
Measure: Number; unit: adverse events
Groups:
- Cohort 1: Target dose of 0.05 X10^8 cells
- Cohort 2: Target dose of 0.4 X10^8 cells
- Cohort 3: Target dose 3.2 x10^8 cells
- Cohort 4: Target dose 26 x10^8 cells
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 5 | 5
adverse events
  Grade 1 Mild | 25 | 19 | 31 | 29
  Grade 2 Moderate | 5 | 9 | 28 | 7
  Grade 3 Severe | 0 | 2 | 6 | 3
  Grade 4 Life Threatening | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants Experiencing Severe or Life Threatening Laboratory Abnormalities
Description: Laboratory measures tested include: hematology, blood chemistry, endocrine values, autoantibodies, and ophthalmologic exam results
  Total number of participants experiencing severe or life-threatening laboratory abnormalities is reported for each cohort. Events reported include hyperglycemia and hypoglycemia.
Time Frame: Mean follow-up of 31 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 5 | 5
Participants
  Any severe or life threatening abnormality | 0 | 1 | 1 | 1
  Abnormality related to study drug | 0 | 0 | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in C-peptide Area Under the Curve
Description: Secondary diabetes-related outcome measure: C-peptide response during mixed meal tolerance test at 26 and 52 weeks, reported as the change from baseline in the area under the curve.
Time Frame: 26 and 52 weeks from baseline
Population: Population includes 14 participants treated.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 4
percentage change from baseline
  26 Weeks | 24.1 (26.6) | 17.4 (19.4) | 14.9 (12.2) | -32.9 (42.9)
  52 Weeks | 25.5 (39.4) | 9.2 (10.2) | -33.9 (6.9) | -48.5 (42.6)

4. Secondary Outcome: Insulin Use
Description: Secondary diabetes-related outcome measure will include insulin use
Time Frame: up to 104 weeks
Population: Population includes 14 participants treated.
Measure: Mean (Standard Deviation); unit: U/day/kg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 4
U/day/kg
  Insulin use at Baseline | 0.127 (0.027) | 0.236 (0.016) | 0.346 (0.211) | 0.298 (0.151)
  Insulin use at Week 26 | 0.193 (0.063) | 0.167 (0.047) | 0.397 (0.080) | 0.294 (0.137)
  Insulin use at Week 52 | 0.245 (0.069) | 0.219 (0.066) | 0.444 (0.108) | 0.385 (0.168)
  Insulin use at Week 104 | 0.334 (0.064) | 0.222 (0.049) | 0.484 (0.050) | 0.550 (0.346)

5. Secondary Outcome: Hemoglobin A1c
Description: Secondary diabetes-related outcome measure will include hemoglobin A1c
Time Frame: Up to 104 weeks
Population: Population includes 14 participants treated
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 4
% of HbA1c
  HbA1c at Baseline | 5.5 (0.8) | 5.6 (0.4) | 6.5 (0.8) | 6.7 (2.2)
  HbAlc at 26 Weeks | 5.5 (0.8) | 5.8 (0.4) | 6.5 (0.9) | 7.2 (2.0)
  HbA1c at 52 Weeks | 6.1 (0.9) | 5.8 (0.6) | 6.7 (1.0) | 7.6 (1.8)
  HbA1c at 104 Weeks | 5.7 (0.8) | 6.1 (0.6) | 6.8 (1.0) | 8.2 (2.3)

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=5) | Cohort 4 (N=5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=5) | Cohort 4 (N=5)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Geographic tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal virus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral ulcers (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Flu like symptoms (General disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 2 (4) | 2 (3) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gluteal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Warts (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (6) | 2 (5) | 4 (9) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Elevated D-dimer (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — left pinky finger
Tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Torn Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Left pectoral muscle
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — bilateral calves-intermittent
Epicondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — right elbow- intermittent
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (4) | 1 (1)
Peripheral sensory nueropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No